CLINICAL TRIAL: NCT00235976
Title: A Multicenter, Randomized, Controlled, Observer-Blinded, Dose-Response Study to Evaluate the Efficacy in Tracheal Intubation and Safety of Gantacurium Chloride for Injection in Healthy Adult Patients Undergoing Surgery With General Anesthesia
Brief Title: The Efficacy and Safety of Gantacurium Chloride for Injection in Tracheal Intubation in Healthy Adult Patients Undergoing Surgery Under General Anesthesia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Avera Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MR/EUM202
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2006-07-21 (Estimated); Status verified 2006-07

CONDITIONS: Healthy
Keywords: Neuromuscular Blocking Agent; Anesthesia; Succinylcholine; Tracheal Intubation; Adjunct for tracheal intubation
MeSH Terms: interventions — Injections

INTERVENTIONS:
Drug: Gantacurium Chloride for Injection (AV430A)

SUMMARY:
This is a multicenter, randomized, controlled, observer-blinded, dose-response study to evaluate the efficacy in tracheal intubation and safety of gantacurium chloride for injection in healthy adult patients undergoing surgery with general anesthesia.

Gantacurium chloride for injection (previously referred to as AV430A) is a new, investigational non-depolarizing ultra-short acting neuromuscular blocking agent (NMB). Preliminary results in animals and healthy human subjects (Phase 1 studies in adult volunteers) suggest that gantacurium chloride for injection may provide a useful adjunct to general anesthesia by permitting rapid intubation. This Phase 2 study will provide more definitive information on the ultra-short acting profile of the compound by determining the quality of intubation in patients, at 60 seconds, as assessed by a blinded intubator. In addition, the safety of the compound will be assessed. In this study, the efficacy and safety of gantacurium chloride for injection will also be compared to a reference drug, succinylcholine, and to placebo.

The primary objective of this study is to determine the dose-response relationship of gantacurium chloride for injection on tracheal intubation conditions after a single rapid bolus intravenous (i.v.) dose as a component of a propofol/opioid induction-intubation sequence and to assess the safety profile of this compound.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between 18 and 65 years of age scheduled for low- or moderate-risk surgical procedure requiring tracheal intubation
* Female patients must not be of child-bearing potential. Females must meet one of the following criteria:

  * Be postmenopausal;
  * Have undergone prior tubal ligation or hysterectomy; or
  * Be scheduled for hysterectomy as the surgical procedure for this study.
* American Society of Anesthesiologists (ASA) Physical Status Classification 1 or 2
* Weight within 30% of ideal body weight
* Able to read and to comprehend information about the study design and procedure; willingness to participate in this study as evidenced by a signed and dated written Informed Consent form
* In good physical and mental health as determined by the procedures/evaluations (completed within 14 days prior to the Induction Phase [scheduled surgical procedure])

Exclusion Criteria:

A patient will not be eligible for inclusion in this study if any of the following criteria are met:

* Evidence of clinically significant cardiovascular, neuromuscular, neurological, psychiatric, renal, hepatic or pulmonary disease (including asthma), or impairment of function (as judged by the investigator)
* Personal or family history of unusual sensitivity to NMBs or other agents used in surgical anesthesia
* Anatomical characteristics recognized as being associated with difficult intubation conditions, even in the presence of complete jaw and vocal cord relaxation
* History or evidence of vocal cord polyps and/or paralysis
* History or evidence of narrow angle glaucoma
* Personal or family history of malignant hyperthermia
* History of major thermal injury that required hospitalization
* Presence of genetically determined disorders of plasma cholinesterase, as determined by medical history
* History or current evidence of abuse of any drug substance, licit or illicit (including alcohol)
* Exposure to any of the following agents within 48 hours prior to the Induction Phase of the study, or, if expected to be administered within the first 15 minutes after administration of study treatment: antibiotics (except penicillins, cephalosporins, and tetracyclines), i.v. lidocaine (except i.v. lidocaine administered in conjunction with propofol to reduce local irritation), quinidine, trimetaphan, or dexamethasone.
* Exposure to any of the following agents within 7 days prior to the Induction Phase of the study: tricyclic antidepressants, phenothiazines, anticonvulsants, antihistamines (H1 - or H2 - receptor antagonists), antihypertensives, antiarrhythmics (including procainamide), beta blockers (including propranolol, calcium channel blockers), diuretics (including furosemide, thiazides, mannitol, and acetazolamide), potent narcotics (including, but not limited to, oxycodone, methadone, morphine, buprenorphine, hydromorphone), and magnesium or lithium salts. Note: weak opioids including, but not limited to, propoxyphene, tramadol, hydrocodone, codeine, meperidine, and tilidine are not reasons for exclusion provided no changes in daily dosage have occurred within 3 days prior to the Induction Phase of the study.
* Exposure to monoamine oxidase inhibitors within 14 days prior to the Induction Phase of the study.
* Exposure to anticholinesterase or cholinomimetic agents within 30 days prior to the Induction Phase
* Previous entry into this or any other study of gantacurium chloride for injection, or participation in any other investigational drug, biologic, or medical device study within 30 days prior to the Induction Phase
* Pregnant (positive pregnancy test during Screening) or breastfeeding/donating breast milk
* Any other condition that, in the opinion of the investigator, would jeopardize the safety or rights of a subject participating in the trial or would render the subject unable to comply with the protocol

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2005-05; Study Completion 2006-03

PRIMARY OUTCOMES:
The primary endpoint in this study is the graded intubation scores at 60 seconds after administration of single rapid i.v. bolus doses of study treatments (gantacurium chloride for injection, succinylcholine, or placebo)

SECONDARY OUTCOMES:
Graded intubation scores at 120 seconds after administration of single rapid i.v. bolus doses of study treatments for those patients in whom the first intubation attempt at 60 seconds failed
Blood pressure (BP) and heart rate (HR) measurements beginning with a propofol/opioid induction-intubation sequence and ending 10 minutes after the initial intubation attempt
12-lead electrocardiograph (ECG) measurements
Number and frequency of adverse events (AEs)
Clinical laboratory data
Vital sign measurements

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Blobner, MD, Principal Investigator — Technischen Universitat Munchen; Jorgen Viby-Mogensen, MD, Principal Investigator — Academic Department of Anasthesia and Intensive Care
Locations (1):
- Technischen Universitat Munchen, Munich, Germany